CLINICAL TRIAL: NCT04624711
Title: A Multicenter, Phase II, Open-label, Single-arm Investigator Initiated Trial to Evaluate the Efficacy and Safety of Eribulin Mesylate Combined With Anlotinib in Metastatic HER2 Negative Breast Cancer Patients
Brief Title: Eribulin Combined With Anlotinib in Metastatic HER2 Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAGER-001
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: HER2-negative Breast Cancer
MeSH Terms: interventions — eribulin; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eribulin Mesylate Combined With Anlotinib (Experimental): Patients receive eribulin mesylate plus anlotinib.
  Interventions: Drug: Eribulin Mesylate; Drug: Anlotinib hydrochloride

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate 1.4mg/m2, administered intravenously on Days 1 and 8 of each 21 day cycle.
  Other Names: Halaven
Drug: Anlotinib hydrochloride — Anlotinib 12mg, administered orally on Days 1-14 of each 21 day cycle.
  Other Names: Anlotinib

SUMMARY:
This is a multicenter, phase II, open-label, single-arm investigator initiated trial to evaluate the efficacy and safety of eribulin mesylate combined with anlotinib in metastatic HER2 negative breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most frequent malignancy in women worldwide. Treatments on metastatic HER2 negative breast cancer are still under exploration. Therefore, it is imperative to find a novel therapy to treat these patients.

This study explores the efficacy and safety of eribulin mesylate combined with anlotinib in metastatic HER2 negative breast cancer patients. The primary objective is to evaluate the progression free survival (PFS). The secondary objective is to evaluate the safety of the combination of eribulin and anlotinib.

ELIGIBILITY:
Inclusion Criteria:

* The patient volunteers and signs an informed consent form;
* Age ≥18 years old, female;
* The patient was diagnosed as HER2 negative breast cancer by histopathology ( HER2 negative (IHC-/+ or IHC++ but FISH/CISH- )), and there is at least 1 measurable lesion of metastasis according to RECIST 1.1;
* All patients have previously underwent chemotherapy containing anthracyclines and taxanes, and received ≥1 line chemotherapy for metastatic breast cancer;
* Patients with hormone receptor positive (ER positive (IHC ER positive percentage ≥1%), PR positive (IHC PR positive percentage ≥1%)) have underwent ≥1 line endocrine therapy;
* Physical condition ECOG PS: 0-1;
* Laboratory tests meet the following criteria:

  1. Bone marrow function: absolute count of blood neutrophils (ANC) ≥1.5×109/L; platelet (PLT)≥100×109/L; hemoglobin (HB)≥90g/L;
  2. Liver function: serum total bilirubin (STB), combined bilirubin (CB) ≤ upper limit of normal (ULN) *1.5; alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN*2.5;
  3. Renal function: serum creatinine (Cr) ≤ ULN; endogenous creatinine clearance (Ccr) ≥ 60 ml / min (calculated using the Cockcroft-Gault formula).

Exclusion Criteria:

* Previous breast cancer history (except for ipsilateral DCIS that only received local treatment ≥5 years ago), malignant tumors of other histological origins (except for non-melanoma skin cancer or cervical carcinoma in situ) unless the patient's tumor had been completely alleviated and had not received treatment for at least 5 years before the enrollment date;
* Major surgery within 4 weeks prior to enrollment, or surgical wounds have not healed;
* Embolization and bleeding occurred within 4 weeks before enrollment;
* Severe cardiovascular disease, including hypertension (BP≥160/95mmHg) uncontrolled by medical treatment, unstable angina, history of myocardial infarction in the past 6 months, congestive heart failure>NYHA II, severe heart rhythm Abnormalities and pericardial effusions;
* Severe infection requires intravenous antibiotic, antifungal or antiviral treatment;
* Other clinical trials of drugs were used in the first four weeks of the first medication;
* Subjects with treatment history of eribulin or anti-angiogenesis drugs;
* Suffering from mental illness, poor compliance;
* Researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 year
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | 2 year
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No